CLINICAL TRIAL: NCT06410664
Title: Safety and Efficiency of the Prolonged (72-hour) Use of a Single Heat and Moisture Exchanger in Adult Mechanically Ventilated Critically Ill and Its Impact on the Lower Respiratory Tract Pathogenic Microbial Colonisation Rate (FILTRex Trial); a Single-centre, Randomised, Controlled Trial
Brief Title: Efficiency and Safety of the Prolonged Use of Heat and Moisture Exchangers in ICU
Acronym: FILTRex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Jiroutková, Kateřina Jiroutková, MD, PhD, DESAIC, Charles University, Czech Republic, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VP/47/0/2022
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: pneumonia; Heat and Moisture Exchange (HME) filter; VAP bundle in ICU; endotracheal tube occlusion
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Intervention Model Description: Eligible patients will be recruited in the medical-surgical ICU at Královské Vinohrady University Hospital (FNKV), managed under an intensivist-led closed ICU, with a 1:1 nurse-to-patient ratio and randomised in equal proportions between HME filter exchange every 72 hours versus daily HME filter exchange arm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, nurses can't be blinded to allocation (the frequency of HME exchange), but are strongly inculcated not to disclose the allocation status of the participant at the follow-up assessments. As the ICU is paperless and fully computerised, the data in the computer can be acquired and analysed by the researchers without having access to information about the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 72-hour HME exchange interval group (Experimental): Intervention group: daily care will be provided according to the local standards, with an HME exchange interval every 72 hours
  Interventions: Other: 72-hour HME exchange interval group
- 24-hour HME exchange interval group (Active Comparator): Control group: daily care will be provided according to the local standards, with an HME exchange interval every 24 hours
  Interventions: Other: 24-hour HME exchange interval group

INTERVENTIONS:
Other: 72-hour HME exchange interval group — All patients in the experimental arm will receive the usual best medical and nursing care with respect to VAP prevention. A dual-limb ventilator circuit with a closed suction system will be used. Bronchodilation or inhalational antibiotics, when ordered, will be delivered by a meshed nebuliser, a part of the ventilatory support circuit and will not be removed between treatments. A closed-circuit suction device will be used, and the frequency of suctioning will be monitored, including the sputum consistency and blood on suctioning. HME filter resistance by estimating the pressure drop over HME using the ventilatory circuit's auxiliary force (Paux) and flow. Temperature and humidity in the ventilator circuit will be measured. HME filters will be exchanged every 72 hours. At the exchange point, both outlets of the HME filter will be swabbed.
  Arms: 72-hour HME exchange interval group
Other: 24-hour HME exchange interval group — All patients in the control arm will receive the usual best medical and nursing care with respect to VAP prevention. A dual-limb ventilator circuit with a closed suction system will be used. Bronchodilation or inhalational antibiotics, when ordered, will be delivered by a meshed nebuliser, a part of the ventilatory support circuit and will not be removed between treatments. A closed-circuit suction device will be used, and the frequency of suctioning will be monitored, including the sputum consistency and blood on suctioning. HME filter resistance by estimating the pressure drop over HME using the ventilatory circuit's auxiliary force (Paux) and flow. Temperature and humidity in the ventilator circuit will be measured. HME filters will be exchanged every 24 hours. At the exchange point, both outlets of the HME filter will be swabbed.
  Arms: 24-hour HME exchange interval group

SUMMARY:
FILTRex is a single-centre, controlled, randomised, prospective, non-inferiority clinical trial to compare the efficiency and safety of prolonged (72-hours) versus standard (24-hours) duration of use for Heat and Moisture Exchange (HME) filters in adult mechanically ventilated critically ill patients

DETAILED DESCRIPTION:
Rationale: Ventilator-associated pneumonia (VAP) is the most common hospital-acquired infection (HAI) in the intensive care unit (ICU), and its impact is very high in terms of morbidity, length of hospital stay and overall costs. Minimising manipulation and disconnection of the ventilator circuit by reducing the frequency of HME filter exchange may lower the risk of its secondary contamination, hence the incidence of VAP, while maintaining its efficacy in terms of sufficient humidification of the inhaled gas mixture and safety in terms of no or minimal change in resistance to airflow.

Aim: To test the effectiveness and safety of prolonged (72-hour exchange interval) use of a single HME.

Design: Prospective, single-centre, parallel-group randomised controlled trial. Subjects: ICU patients (general ICU)

Treatment in the intervention group: HME filter exchange every 72 hours

Control group: Standard-of-care: daily HME filter exchange

Primary outcome:

1. Presence of HME-associated adverse events (a composite endpoint of endotracheal tube occlusion or nosocomial tracheobronchitis or pneumonia).
2. The cumulative incidence of lower respiratory tract microbial colonisation analysed by the Kaplan-Maier method, censored in the case of ICU discharge or extubation > 24h.

Secondary and exploratory outcomes: Differences in the relative risk of infection-related ventilator-associated complications, antibiotics (ATB) exposure analysis, length of ICU stay in days (time frame: three months), number of ventilator-free days (time frame: 28 days); differences in the incidence of endotracheal tube occlusion necessitating reintubation between individual groups, differences in airway resistance, humidity delivered to the patients and efficacy of HMEs between groups

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. In-patient in ICU and expected to stay > 3 days
3. Mechanical ventilation or imminent need of it; predicted length of mechanical ventilation ≥ 72h
4. Clinical Pulmonary Infection score (CPIS) less than six at the baseline 5 No history and symptoms of aspiration at the baseline

Exclusion Criteria:

1. Suspected pulmonary infection on admission and in the first 48 hours of mechanical ventilation
2. Pregnancy
3. Acute respiratory distress syndrome
4. Body temperature < 32°C
5. Airway bleeding or other contraindications for the use of HME
6. An early decision of treatment withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence of HME-associated adverse events | 3 months
  A composite endpoint of nosocomial tracheobronchitis or pneumonia (all-cause, nosocomial and ventilator-associated) or endotracheal tube occlusion).
The cumulative incidence of lower respiratory tract microbial colonisation analysed by the Kaplan-Maier method, censored in the case of ICU discharge or extubation > 24h. | 3 months
  To detect microorganisms in the lower respiratory tract, tracheal aspirate will be directly cultured for detecting Gram-positive, Gram-negative, and anaerobic bacteria and fungi. Standard microbial surveillance (tracheal aspirate) will be performed on admission, twice a week (Monday, Thursday) and always ad hoc according to the clinical situation.

SECONDARY OUTCOMES:
Differences in the relative risk of infection-related ventilator-associated complications (IVAC) according to the Centers for Disease Control and Prevention (CDC) criteria. | 3 months
  Incidence rates among patients exposed to experimental intervention compared to those receiving standard care. We will establish the IVAC diagnosis based on the following:
  * an increase of the daily minimum positive end-expiratory pressure (PEEP) of ≥3 cm of water column (H2O) and (or) the daily minimum inspired oxygen fraction (FiO2) of ≥20 points sustained for ≥2 days and
  * evidence of a new infection present (abnormal temperature or white blood cell count) and prescription of a new antibiotic for ≥4 days
ATB exposure analysis | 3 months
  Duration of antibiotics prescribed at discharge.
Length of ICU stay in days | 3 months
  that is, length in ICU stay in days
Number of ventilator-free days. | at 28 days
  That is, the number of days, out of 28 days after admission, that the patient has not been supported by mechanical ventilation.

OTHER OUTCOMES:
The length of ATB therapy until extubation, death or IVAC. | 3 months
  Cumulative percentage of days on the ventilator with ATB until extubation, death or IVAC.
The values of HME performance in vivo (temperature) during mechanical ventilation. | up to 30 days
  The absolute temperature of input, load, return, loss, yield, and thermal differential, their variation over time (72 hours) and the differences between in vivo obtained values of HME performance indicators and their laboratory values declared by the manufacturer in the technical sheet and prescribed by the international standard.
The values of HME performance in vivo (humidity) during mechanical ventilation. | up to 30 days
  The absolute humidity of input, load, return, loss, yield, and thermal differential, their variation over time (72 hours) and the differences between in vivo obtained values of HME performance indicators and their laboratory values declared by the manufacturer in the technical sheet and prescribed by the international standard.
The change in resistance of the HME filter from day 0 to day 2 (72 hours) and during drug nebulisation | up to 30days
  The pressure drops over HME filter during mechanical ventilation.
The change in resistance of the HME filter during drug nebulisation | up to 30 days
  The pressure drop over HME filter during drug nebulisation.

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Jiroutková, Principal Investigator — 3rd Faculty of Medicine, Charles University and FNKV, Prague
Locations (1):
- 3rd Faculty of Medicine and FNKV, Prague, Česká Republika, Czechia